CLINICAL TRIAL: NCT04311333
Title: Endostomal Three-dimensional Ultrasonography Compared to Clinical Examination, Computerized Tomography and Intraoperative Findings for Parastomal Hernia Diagnosis
Brief Title: Endostomal Three-dimensional Ultrasonography for Parastomal Hernia
Acronym: CTULOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTULOP
Record Dates: First submitted 2020-03-12; First posted 2020-03-17 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Parastomal Hernia
Keywords: Parastomal hernia; Ultrasound; Ultrasonography; Endostomal; Intrastomal; Colostomy; Ileostomy
MeSH Terms: interventions — Physical Examination; Laparoscopy

STUDY DESIGN:
Intervention Model Description: All patients will be examined with endostomal three-dimensional ultrasonography, clinical examination and computerized tomography before undergoing laparotomy or laparoscopy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): All patients undergo endostomal three-dimensional ultrasonography, computerized tomography, clinical examination and laparotomy/laparoscopy.
  At all the respective examinations, the presence of a parastomal hernia as well as hernia location and size is evaluated.
  Interventions: Diagnostic Test: Endostomal three-dimensional ultrasonography; Diagnostic Test: Computerized tomography of the abdomen; Diagnostic Test: Clinical examination; Diagnostic Test: Evaluation at laparotomy/laparoscopy

INTERVENTIONS:
Diagnostic Test: Endostomal three-dimensional ultrasonography — Examination with rectal probe enclosed by water-filled balloon. Rectal mode. Dynamic examination in different positions with and without increased intra-abdominal pressure.
Diagnostic Test: Computerized tomography of the abdomen — Supine position, without increased intra-abdominal pressure. Experienced radiologist interprets the examination.
  If adequate examination has already been performed within the last 10 months, these images will be used and the patient will thus not undergo computerized tomography within the study.
Diagnostic Test: Clinical examination — Patients will be clinically examined with inspection and palpation in supine and erect position with and without increased intra-abdominal pressure.
Diagnostic Test: Evaluation at laparotomy/laparoscopy — During laparotomy or laparoscopy, inspection and/or palpation of the stoma at the abdominal wall orifice is performed.

SUMMARY:
The intention is to examine the role of ultrasonographic examination inside intestinal stomas in diagnosing parastomal hernia. Patients with a stoma since at least one year back who are being scheduled for abdominal surgery will be examined for eligibility according to the selection criteria. Included patients will undergo routine clinical examination, endostomal ultrasonography and computerized tomography scan of the abdomen. Findings will be correlated to findings during surgery (gold standard). Values for sensitivity, specificity, predictive values and likelihood ratio will be calculated.

DETAILED DESCRIPTION:
Parastomal hernia (PSH) is one of the most common stoma complications, with an incidence of 30-50 % within just a couple of years of stoma creation. Surgical parastomal hernia repair is a morbid and complicated procedure, with a 30-day reoperation rate of 13 % and 30-day mortality rate of 6 % in population-based surveys. There is no established gold standard diagnostic modality. Routinely, patients are examined clinically in various positions with and without increased intra-abdominal pressure. It has been shown in previous studies that clinical examination has a very low inter-observer reliability. Computerized tomography is often performed in addition to clinical examination, but is not ideal in diagnosing PSH either, not only beacause of insufficient test characteristics but also since the examinations should ideally be performed with specific protocols, prone position and be reviewed by a dedicated radiologist. The risk of incorrectly diagnosing a PSH (false positive) is that patients might subsequently be exposed to complex and dangerous surgical interventions without any health benefit, while incorrectly ruling out a PSH (false negative) can cause the patient to have to live with potentially treatable symptoms, life-threatening bowel incarceration being the most severe potential complication.

Thus, improved diagnostic accuracy is required. A method that has been developed within our research group is endostomal tree-dimensional ultrasonography, which has preliminarily proven to be approximately as sensitive as CT, with a markedly higher specificity. A larger and less selected study needs to be conducted in order to reliably calculate test characteristics, predictive values and likelihood ratio.

ELIGIBILITY:
Inclusion Criteria:

* End colostomy or end ileostomy since ≥ 1 year
* Planned for laparotomy or laparoscopy
* Age ≥ 18
* Speaks and reads Swedish language
* Informed consent

Exclusion Criteria:

* Known parastomal hernia only indication for laparotomy or laparoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-09-27 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Test characteristics | ≥ 1 year since stoma creation
  Sensitivity, specificity, predictive values, likelihood ratio

CONTACTS AND LOCATIONS:
Overall Officials: Karin Strigård, Principal Investigator — Department of Surgical and Perioperative Sciences, Umeå University
Locations (3):
- Sweden (3):
  - Sunderby Hospital, Luleå, Norrbotten County
  - Södertälje Hospital, Södertälje, Stockholm County
  - University Hospital of Umeå, Umeå, Västerbotten County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gurmu A, Matthiessen P, Nilsson S, Pahlman L, Rutegard J, Gunnarsson U. The inter-observer reliability is very low at clinical examination of parastomal hernia. Int J Colorectal Dis. 2011 Jan;26(1):89-95. doi: 10.1007/s00384-010-1050-2. Epub 2010 Sep 7. PMID 20821218
- [Background] Gurmu A, Gunnarsson U, Strigard K. Imaging of parastomal hernia using three-dimensional intrastomal ultrasonography. Br J Surg. 2011 Jul;98(7):1026-9. doi: 10.1002/bjs.7505. Epub 2011 Apr 20. PMID 21509751
- [Background] Strigard K, Gurmu A, Nasvall P, Pahlman P, Gunnarsson U. Intrastomal 3D ultrasound; an inter- and intra-observer evaluation. Int J Colorectal Dis. 2013 Jan;28(1):43-7. doi: 10.1007/s00384-012-1526-3. Epub 2012 Jul 7. PMID 22772711
- [Background] Nasvall P, Wikner F, Gunnarsson U, Rutegard J, Strigard K. A comparison between intrastomal 3D ultrasonography, CT scanning and findings at surgery in patients with stomal complaints. Int J Colorectal Dis. 2014 Oct;29(10):1263-6. doi: 10.1007/s00384-014-1944-5. Epub 2014 Jul 2. PMID 24986139